CLINICAL TRIAL: NCT06211582
Title: Clinical Performances of 3-different Tooth-colored Restorative Materials in Class-II Cavities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Kemal Işıklı, Principal Investigator, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA-22015
Record Dates: First submitted 2024-01-09; First posted 2024-01-18 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Caries,Dental
Keywords: Alkasite-based; Posterior resin composite; Class II restoration; Glass Hybrid
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cention N (Ivoclar Vivadent, Schaan, Liechtenstein) (Experimental): Powder: Calcium-fluoro-silicate glass, barium glass, calcium-barium-aluminium fluoro-silicate glass, iso-fillers, ytterbium trifluoride, initiators and pigments. Liquid: Dimethacrylates, initiators, stabilizers, additives and mint flavour. The mixing ratio was 2 parts powder and 2 drops of liquid or 3 parts powder and 3 drops.After distributing the powder and liquid side by side on a mixing pad, the liquid was spread to expand the surface.The first part of the powder was mixed with the entire liquid dispensed on the mixing pad.After the components have been thoroughly mixed, add the remaining powder and stirred again until a homogeneous consistency is obtained (45 - 60 seconds). After careful adaptation to the cavity and densification, occlusal excesses were removed.
  Interventions: Device: Cention N (Ivoclar Vivadent, Schaan, Liechtenstein)
- Equia Forte HT ( GC, Tokyo, Japan) (Experimental): Powder: 95% strontium fluoroalumino-silicate glass. Liquid: 5% polyacrilic acid.
  Equia Forte HT was mixed in a capsule (10 seconds) and injected into the cavity. After a 2.5 min curing time, occlusal excesses were removed. Equia Coat (GC, Tokyo, Japan) was then applied and light-cured (D-Light Pro, GC, Tokyo, Japan 1,400 mW/cm2) for 20 seconds.
  Interventions: Device: Equia Forte HT ( GC, Tokyo, Japan)
- Gradia Direct Posterior ( GC, Tokyo, Japan) (Experimental): Matrix: Urethanedimethacrylate (UDMA), dymethacrylate camphorquinone. Filler: fluoro-alumino-silicate glass silica powder.
  After completing the cavity, the enamel surface was selectively roughened using 37% orthophosphoric acid for 30 seconds. Subsequently, GC Solare Universal Bond adhesive agent (GC Corp., Tokyo, Japan) was utilized. It was applied in 2mm layers in accordance with the composite manufacturer's instructions. Each layer was polymerized for 20 seconds.
  Interventions: Device: Gradia Direct Posterior ( GC, Tokyo, Japan)

INTERVENTIONS:
Device: Cention N (Ivoclar Vivadent, Schaan, Liechtenstein) — The Alkasite-Based Tooth-Colored Material
  Arms: Cention N (Ivoclar Vivadent, Schaan, Liechtenstein)
Device: Equia Forte HT ( GC, Tokyo, Japan) — Glass Hybrid Restorative Material
  Arms: Equia Forte HT ( GC, Tokyo, Japan)
Device: Gradia Direct Posterior ( GC, Tokyo, Japan) — Conventional Composite Resin
  Arms: Gradia Direct Posterior ( GC, Tokyo, Japan)

SUMMARY:
The goal of this clinical trial comparatively investigate the clinical performances of 3 different tooth-colored restorative materials in the treatment of Class II cavities after 6 months and one year.

DETAILED DESCRIPTION:
High plaque accumulation at the proximal surfaces of posterior teeth can lead to the development of caries and the necessity of dental treatments.The complexity of application methods for resin composites could influence the risk of secondary caries due to bacterial microleakage.In modern dentistry, simplified, esthetic, and satisfactory restoration of tooth decay has led to innovative material developments.Rapidly cured restorative materials applied in large increments with self-adhesive properties became an important solution for easy and effective applications.

Restorative materials with bioactive or caries-protective abilities have been introduced, such as glass hybrid materials. Recently, to overcome the limitations of restorative materials, it was attempted to add caries-protective ions, especially alkaline and alkaline earth ions, such as calcium, in addition to phosphate or fluoride. This newly introduced material contains alkalizing properties due to the release of hydroxyl ions.

In 2016, Ivoclar Vivadent developed a new restorative material consisting of a powder and a liquid part and commercially named this product "Cention N".

Cention N has bioactive properties like glass ionomer cements. It has been developed to prevent demineralisation by neutralising acids through ion release. It contains alkaline fillers. Therefore, a new classification as "Alkasites" has emerged.

One lesion in each patient will be randomly assigned to be restored using either the GC Gradia Direct Posterior, Cention N and Equia Forte HT. The adhesive, GC Solare Universal Bond will be used for adhesive procedures. The clinical procedure for the restorations will be performed by a single operator. The restorations will be evaluated by two calibrated examiners at baseline and at 6, 12, months in accordance with the FDI criteria. Data will be statistically analyzed using the Chi-square and Fischer's exact tests (p < 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals who do not have any systemic disease that prevents restorative treatment
* Individuals between the ages of 18-65
* Brushing your teeth twice a day
* Having at least 20 teeth in occlusion and at least 3 approximal lesions with antagonist teeth in the opposite arch
* Volunteer individuals who agree to participate in the research and sign the informed consent form and who have undergone initial periodontal treatment will be included in the study.

Exclusion Criteria:

* Pregnant or breastfeeding women
* Individuals with advanced periodontal disease
* Individuals using removable partial dentures
* Individuals with bruxism
* Individuals with malocclusion
* Patients with known allergies to resin-based restorative materials and bonding agents
* Patients with a history of allergy to local anesthesia
* Endodontic treatment, teeth that need pulp capping or endodontic treatment is available

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2022-08-28 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Surface gloss/lustre and roughness | From Baseline to 12 Month
  Observers evaluated the restorations was performed using FDI criteria regarding surface gloss/lustre and roughness. Surface gloss/lustre and roughness was evaluated by 2 independent clinicians. Visual inspection with a mirror was performed.Scores; 1: Comparable to enamel 2: Slightly dull, not noticeable from speaking distance 3: Dull surface but acceptable if covered with film of saliva 4: Rough surface, cannot be masked by saliva film, simple polishing is not sufficient 5: Quite rough, unacceptable plaque retentive surface
Surface and marginal staining | From Baseline to 12 Month
  Observers evaluated the restorations was performed using FDI criteria regarding surface and marginal staining. Surface and marginal staining was evaluated by 2 independent clinicians. Visual inspection with a mirror was performed. Scores; 1: No marginal or surface staining 2: . Minor staining, easily removable 3: Moderate staining not noticeable from a speaking distance, also present on other teeth. Not aesthetically unacceptable 4: Surface staining recognizable from speaking distance. Or severe localized marginal staining not removable by polishing 5: Severe surface staining or unacceptable. Generalized and profound marginal discoloration.
Colour match/stability and translucency | From Baseline to 12 Month
  Observers evaluated the restorations was performed using FDI criteria regarding colour match/stability and translucency. Colour match/stability and translucency was evaluated by 2 independent clinicians. Visual inspection with a mirror was performed. Scores; 1: Colour and translucency of the restoration have a clinically excellent match with the surrounding enamel 2: Minor deviations in shade between tooth and restoration are apparent 3: Clear deviation but acceptable. Does not affect aesthetics 4: Colour and/ or translucency are clinically unsatisfactory, recognisable from speaking distance 5: Colour match and/or translucency are clinically unsatisfactory
Anatomic form | From Baseline to 12 Month
  Observers evaluated the restorations was performed using FDI criteria regarding anatomic form. Anatomic form was evaluated by 2 independent clinicians. Visual inspection with a mirror was performed. Scores; 1: Form is ideal 2: Form deviates slightly from the remainder of the tooth 3: Form differs but is not aesthetically displeasing 4: Anatomic form is altered, the aesthetic result is unacceptable 5: Anatomic form is unsatisfactory and/or lost
Fracture of restorative material and retention | From Baseline to 12 Month
  Observers evaluated the restorations was performed using FDI criteria regarding fracture of restorative material and retention. Fracture of restorative material and retention was evaluated by 2 independent clinicians. Visual inspection with a mirror was performed. Scores; 1: Restoration retained, no fractures, cracks or chipping 2: Small hairline crack 3: Two or more or larger hairline cracks and/or chipping (not affecting the marginal integrity or proximal contact) 4: Chipping fractures affect marginal quality and/or proximal contacts; bulk fractures with or without partial loss of (<1/2 of the restoration) 5: (Partial or complete) loss of the restoration
Marginal adaptation | From Baseline to 12 Month
  Observers evaluated the restorations was performed using FDI criteria regarding marginal adaptation. Marginal adaptation was evaluated by 2 independent clinicians. Visual inspection with a mirror was performed. Scores; 1: Harmonious outline, no gaps, no discoloration 2: Small marginal chip fracture can be eliminated by polishing 3: Vertical/horizontal gap <250 μm, easily perceptible with a blunt explorer with a tip diameter of 250 μm. Several small marginal fractures cannot be modified without damage and are unlikely to cause longterm effects 4: Vertical/horizontal gap > 250 μm, may result in exposure of dentine or base 5: Restoration is loose but in situ
Proximal contact point and food impaction | From Baseline to 12 Month
  Observers evaluated the restorations was performed using FDI criteria regarding proximal contact point and food impaction. Proximal contact point and food impaction was evaluated by 2 independent clinicians. Visual inspection with a dental floss and metal blades was performed. Scores; 1: Normal contact point (dental floss can be inserted but not 50 μm blade) 2: Slightly too strong but acceptable. Floss can only be passed with force 3: Slightly too weak (50 μm metal blade can pass easily whereas 100 μm [two blades] cannot) 4: 100 μm (two 50 μm metal blades) can easily pass and possible damage (food impaction) 5: Too weak and/ or clear damage (food impaction) and/or pain gingivitis
Radiographic examination | From Baseline to 12 Month
  Observers evaluated the restorations was performed using FDI criteria regarding radiographic examination. Radiographic examination was evaluated by 2 independent clinicians.Scores; 1: No pathology, harmonious transition between restoration and tooth 2: Small visible but acceptable excess and/or a positive/ negative step or gap <150 μm 3: Gaps and/or positive/negative step <250 μm 4: Gaps and/or positive/negative step >250 μm and/or marked interradicular excess material 5: Gaps >500 μm and/ or secondary caries or apical pathology, tooth/ restoration fracture
Postoperative sensitivity and tooth vitality | From Baseline to 12 Month
  Observers evaluated the restorations was performed using FDI criteria regarding postoperative sensitivity and tooth vitality. Postoperative sensitivity and tooth vitality was evaluated by 2 independent clinicians. Scores; 1: No hypersensitivity, normal vitality 2: Low hypersensitivity for a limited period of time, normal vitality 3: Premature/slightly more intense or delayed/weak hypersensitivity. No subjective complaints 4:Premature/very intense or extremely delayed/weak hypersensitivity with subjective complaints. Or negative sensitivity 5: Very intense, acute pulpitis or non vital tooth. Removal of restoration with or without immediate root canal treatment is required or the tooth must be extracted
Recurrence of initial pathology (secondary caries) | From Baseline to 12 Month
  Observers evaluated the restorations was performed using FDI criteria regarding recurrence of initial pathology (secondary caries). Recurrence of initial pathology (secondary caries) was evaluated by 2 independent clinicians. Visual inspection with a mirror was performed. Scores; 1: No secondary or primary caries 2: Very small, localized demineralization area 3: Larger areas of demineralisation, preventive measures necessary (dentine not exposed) 4: Caries with cavitation 5: Deep secondary caries or exposed dentine that is not accessible for repair
Tooth cracks and fractures | From Baseline to 12 Month
  Observers evaluated the restorations was performed using FDI criteria regarding tooth cracks and fractures. Tooth cracks and fractures was evaluated by 2 independent clinicians. Visual inspection with a mirror was performed. Scores; 1: Complete integrity 2: Minor marginal crack or a hairline crack which cannot be probed. The patient has no clinical symptoms 3: Enamel split or crack <250 μm. No adverse effects 4: Major enamel split (gap >250 μm or dentine/base exposed. Or crack>250 μm (explorer penetrates) 5: Cusp or tooth fracture
Localised reactions of soft tissue | From Baseline to 12 Month
  Observers evaluated the restorations was performed using FDI criteria regarding localised reactions of soft tissue. Localised reactions of soft tissue in direct contact with the restoration was evaluated by 2 independent clinicians. Scores; 1: Healthy mucosa adjacent to restoration 2: Healthy after minor removal of mechanical irritations (sharp edges etc.) 3: Alteration of mucosa but no suspicion of causal relationship with filling material 4: Suspected mild allergic, lichenoid or toxicological reaction 5: Suspected severe allergic, lichenoid or toxicological reaction
Oral and somatic/ psychiatric symptoms | From Baseline to 12 Month
  Observers evaluated the restorations was performed using FDI criteria regarding oral and somatic/ psychiatric symptoms. Oral and somatic/ psychiatric symptoms in direct contact with the restoration was evaluated by 2 independent clinicians. Scores; 1: No symptoms of adverse effects 2: Short-term minor transient symptoms 3: Minor oral and/or general symptoms of malaise 4: Persistent oral/general symptoms, recurrent symptoms 5: Acute/severe oral/general symptoms requires immediate replacement

CONTACTS AND LOCATIONS:
Overall Officials: Filiz Yalçın Çakır, Prof., Principal Investigator — Hacettepe University; Uzay Koç Vural, Assoc. Prof., Principal Investigator — Hacettepe University; Kemal Işıklı, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Gurgan S, Kutuk ZB, Yalcin Cakir F, Ergin E. A randomized controlled 10 years follow up of a glass ionomer restorative material in class I and class II cavities. J Dent. 2020 Mar;94:103175. doi: 10.1016/j.jdent.2019.07.013. Epub 2019 Jul 25. PMID 31351909
- [Result] Bektas Donmez S, Uysal S, Dolgun A, Turgut MD. Clinical performance of aesthetic restorative materials in primary teeth according to the FDI criteria. Eur J Paediatr Dent. 2016 Sep;17(3):202-212. PMID 27759409
- See also: Related info — https://www.gc.dental/europe/en/products/equiaforteht
- See also: Related info — https://www.gc.dental/europe/en/products/gradiadirect
- See also: Related info — https://www.ivoclar.com/en_us/eifu?document-id=36696&show-detail=1